Prognostic value of the levels of circulating tumor cells (CTCs) in peripheral blood in patients with prostate cancer at high risk (Clinical Stages IIB-III) treated radically with radiotherapy and hormone therapy

Unique Protocol ID: CaPr-RTCTC-01/PI 197 Version 2, October 10<sup>th</sup> 2012

NTC01800058

Almudena Zapatero MD, PhD – Radiation Oncology Department
HOSPITAL UNIVERSITARIO DE LA PRINCESA

Prognostic value of the levels of circulating tumor cells (CTCs) in peripheral blood in patients with prostate cancer at high risk (Clinical Stages IIB-III) treated radically with radiotherapy and hormone therapy.

# **HYPOTHESIS:**

The detection and quantification of Circulating tumor cells CTCs in peripheral blood of patients with prostate adenocarcinoma may be useful at least for:

- Getting a correct stratification of patients with high-risk prostate cancer (PCa).
- Set the prognosis at baseline.
- Evaluate the response to different treatments (predictive value and monitoring).
- Establish individualized therapies.

## **MAIN AIM:**

Primary Objective:

To evaluate the proportion of patients with high-risk prostate cancer (NCCN 2011), IIB-III AJCC staging, that expresses circulating prostatic tumor cells (CTCs) in the peripheral blood (PB).

#### **SECONDARY AIMS:**

To establish whether the expression of CTCs a) following neoadjuvant androgen deprivation (AD) prior to radiotherapy (RT) and b) following RT, predict for biochemical relapse, overall survival and distant metastasis.

#### **METHODOLOGY:**

Prospective analysis of biologic samples from peripheral blood of 65 patients with localized high-risk PCa (NCCN 2011) treated with RTC-3D-IMRT combined with AD.

Following the sign of the informed consent of the patient, the blood samples will be analyzed for CTCs using an immunomagnetic method based on the CellSearch system (Veridex), in 3 periods of time:

- a) prior to any treatment;
- b) Following AD and prior to RT; and
- c) Following the end of RT (1-3 months afterwards).

4) 6-12 months following the end of RT in those patients with 0 CTCs in the first determination and positive CTCs in the following determinations. A cut off of 0 vs ≥ 1CTCs/7.5 mL blood was defined as a threshold for negative versus positive CTCs status.

Comparison between the expression of CTCs in peripheral blood before and following AD and RT will be performed. The quantification of the CTCs obtained in these phases of treatment will be correlated with the treatment results in terms of biochemical failure according to Phoenix definition, distant metastasis rate and overall survival to identify a significant prognostic relationship and to determine the potential effect of the treatment in the number of CTCs

Our working group will include 65 patients because the amount is based on routine clinical activity can be safely enrolled in the project development time by the participating centers.

# **NUMBER OF PATIENTS:**

65 patients

## **CONDITION:**

This research project will take place in the context of clinical practice, without the need of complementary extras or additional visits. Treatment given standard treatment is recommended in clinical practice guidelines. Finally, the extraction of 7.5 ml of blood needed will be in the same procedure as usual veno-puncture for clinical testing for the diagnosis and monitoring of patients.

After obtaining informed consent shall be the removal of SP samples (7.5 ml) for detection of CTCs by immunomagnetic method based on the CellSearch system (Veridex) in three time periods:

- a) Prior to the start of any treatment-DA initially neoadjuvant
- b) Prior to the start of RT (DA after neoadjuvant)
- c) At the end of RT (1-3 months)

The analysis-quantification of CTCs obtained in these phases, will correlate with treatment outcomes in terms of biochemical failure (BF) according to the criteria of Phoenix 2006 and overall survival to identify potential prognostic value. Likewise determinations are compared before and after CTCs DA and RT to evaluate the effect of such treatments on modular quantifying CTCs

The assignment of a patient to a particular therapeutic strategy is independent prior to the decision to include the patient in the study. The study period is after the start of the investigation.

# **INTERVENTION:**

This is a multicenter, prospective, observational, single-arm, phase IV.

Prospective analysis of biological material from samples of peripheral blood (PB) of patients diagnosed with prostate cancer at high risk (NCCN 2011), AJCC stage IIB-III, treated with 3D-CRT, IMRT dose escalation (with androgen deprivation (DA))

After obtaining informed consent shall be the sampling of peripheral blood (PB) for detection of CTCs in three treatment periods:

- Before starting any treatment-DA initially neoadjuvant
- Prior to the start of RT (DA after neoadjuvant)
- At the end of RT (1-3 months)

The analysis-quantification of CTCs obtained in these phases, will correlate with treatment outcomes in terms of biochemical failure (BF) according to the criteria of Phoenix 2006 and overall survival and metastasis-free to identify potential prognostic value. Likewise determinations are compared before and after CTCs DA and RT to evaluate the effect of such treatments on modular quantifying CTCs (predictive value).

## PHASE:

A multicenter, prospective, observational, single-arm, phase IV.

## STUDY TYPE: STUDY DESIGN:

A multicenter, prospective, observational, single-arm, phase IV.

Prospective analysis of biological material from samples of peripheral blood (PB) of 65 patients diagnosed with prostate cancer at high risk (NCCN 2011), AJCC stage IIB-III, treated with 3D-CRT, IMRT dose escalation and androgen deprivation (DA).

# **OFFICIAL TITLE:**

Prognostic value of the levels of circulating tumor cells (CTCs) in peripheral blood in patients with prostate cancer at high risk (Clinical Stages IIB-III) treated radically with radiotherapy and hormone therapy. " Ref.: CaPr-RTCTC-01/PI 197

## PRIMARY OUTCOME MEASURE:

The expression of circulating tumor cells in the peripheral blood of patients with high-risk prostate cancer (NCCN 2011) (Initially a cutoff point of  $\square$  3 or more circulating cells per 7.5 ml of blood will be taken as the reference baseline).

## **SECUNDARY OUTCOME MEASURES:**

- Radiation dose
- Duration and type of hormone therapy
- Gleason sum
- Pretreatment PSA
- Clinical T stage
- Biochemical failure-free survival ("Phoenix definition": PSA ≥ 2 ng/ml over the nadir PSA).
- Overall Survival defined as death due to any cause
- Metastasis-free survival defined as imaging documented evidence of distant spread of disease;

## **ARMS**:

Not applicable

## **ASSIGNED INTERVENTIONS:**

The experimental approximations that will be develop in this project are enumerated below:

Patients that satisfy inclusion criteria, and after signing informed consent, will extract 1 blood sample (7.5 mL):

- a) prior to any treatment;
- b) Following AD and prior to RT; and
- c) Following the end of RT (1-3 months afterwards).
- 4) 6-12 months following the end of RT in those patients with 0 CTCs in the first determination and positive CTCs in the following determinations. A cut off of 0 vs ≥ 1CTCs/7.5 mL blood was defined as a threshold for negative versus positive CTCs status.

The quantification of CTC in blood samples will be done with the CellSearch® system.

#### **ELIGIBILITY**:

#### AGES ELIGIBLE FOR STUDY:

Patients aged > 18

#### **GENDERS ELIGIBLE FOR STUDY:**

Male

# **INCLUSION CRITERIA:**

- Patients aged > 18 with capacity to give informed consent.
- Patients with histologically confirmed prostate cancer.
- Patients with a high risk factor: PSA> 20 ng / ml, Gleason 8-10 and / or stage T3a-b, N0M0 (NCCN 2011, stage IIB-III AJCC classification 2010).
   Staging by: Histology-Gleason score-, PSA, TR, ECO TR, CT, MRI.
- Patients who accept radical treatment with radiotherapy.
- Patients who give written informed consent to participate in the study.

# **EXCLUSION CRITERIA:**

- a) Any patient diagnosed with prostate cancer, which does not meet the prerequisites.
- b) Any patients with another malignancy diagnosed in the past 5 years (except basal cell or squamous cell carcinoma of skin).
- c) Any patient who has prostate biopsy performed 7 days prior to study entry.
- d) Patients who have received prior treatment with hormonal therapy, chemotherapy or radiotherapy.
- e) Patients with PSA> 100 ng / ml.
- f) Any situation or condition of the patient which in the opinion of the investigator, advised against participation in the study.

#### STATISTICAL METHODS

The frequency of expression of CTCs was estimated with its 95% confidence interval (CI). Initially a cutoff point of ≥3 CTCs/7.5 mL of blood was taken as the

reference baseline. Because of the low CTC counts observed and for statistical purposes, we empirically established a cut-off of 0 vs  $\geq$ 1 CTCs/7.5 mL blood as the thresholds between negative and positive CTC status. The association between the presence and development of CTCs over time and well-known clinicopathological features was assessed using the  $\square$ 2 test or Fisher exact test. Overall survival, metastasis-free survival, and biochemical failure—free survival were estimated using the Kaplan-Meier method. The curves were compared using the log-rank test. All events were defined as time until death from any cause (OS), distant metastasis (MFS), biochemical failure (bFS), or date of last follow-up visit. Cox regression models were constructed to estimate the hazard ratio and 95% CI as a measure of the effect and were adjusted for potential confounding variables (P  $\leq$  0.20)..All hypothesis tests were performed using 2-tailed alternatives. Statistical significance was set at P < 0.05.

# **CONTACTS AND LOCATION:**

Almudena Zapatero, MD PhD, IP

Hospital Universitario de la Princesa

Radiation Oncology Department

C/Diego de León, 62

Madrid 28006

E-mail: azapatero.hlpr@salud.madrid.org

## **PUBLICATIONS:**

- 1. D'Ambert JE. Prostate cancer. Lancet 2008; 371:1710-21
- 2. Zelefsky MJ, Yamada Y, Fuks Z, et al. Long-term results of conformal radiotherapy for prostate cancer: Impact of dose escalation on biochemical tumor control and distant metastases-free survival outcomes. Int J Radiat Oncol Biol Phys 2008;71:1028–1033.
- 3. KubanDA, Tucker SL, Dong YL, et al. Long-term results of the M.D. Anderson randomized dose-escalation trial for prostate cancer. Int J Radiat Oncol Biol Phys 2008;70:67–74.
- 4. Roach M 3rd, Bae K, Speight J, et al. Short-term neoadjuvant androgen deprivation therapy and external-beam radiotherapy for locally advanced prostate cancer: Long-term results of RTOG 8610. J Clin Oncol 2008;26:585–591.
- 5. Bolla M, Collette L, Van Tienhoven G, et al. Ten-year results of long-term adjuvant androgen deprivation with goserelin in patients with locally advanced prostate cancer treated with radiotherapy: A phase III EORTC study. Int J Radiat Oncol Biol Phys 2008;72:S30–S31.
- 6. Horwitz EM, Bae K, Hanks GE, et al. Ten-year follow-up of Radiation Therapy Oncology Group protocol 92-02: A phase III trial of the duration of

- elective androgen deprivation in locally advanced prostate cancer. J Clin Oncol 2008;26:2497–2504.
- 7. A. Cabanes, E. Vidal, N. Aragones, B. Perez-Gomez, M. Pollan, V. Lope et al. Cancer mortality trends in Spain: 1980–2007. Annals of Oncology 21 (Supplement 3): iii14–iii20, 2010.
- 8. L. Resel Folkersma, C. Olivier Gómez, L. San José Manso, et al. Cuantificación Inmunomagnética De Células Tumorales Circulantes En Pacientes Con Cáncer De Próstata: Correlación Clínica Y Patológica. Arch. Esp. Urol. 2010; 63 (1): 23-31
- 9. Ghossein RA, Bhattacharya S and Rosai J. Molecular detection of micrometastases and circulating tumor cells in solid tumors. Cin Cancer Res 1999; 5:1950-60.
- 10. Llanes L, Ferruelo A, Lujan M, et aol. Quantitative real-time reverse transcription: polymerase chain reaction of prostate-specific antigen for detection of circulating prostatic cells in patients with clinically localized prostate cancer. Prostate Cancer and Prostatic diseases 2005; 8:248-52.
- 11. A Zapatero, F Valcárcel, F A Calvo, et al. Risk-adapted androgen deprivation and escalated 3D-Conformal radiotherapy for prostate cancer: Does radiation dose influence outcome of patients treated with adjuvant androgen deprivation? Report of a multicenter trial (GICOR 05/99). J Clin Oncol 2005;23:6561-6568.
- 12. Roach M III, Hanks G, Thames H Jr., et al. Defining biochemical failure following radiotherapy with or without hormonal therapy in men with clinically localized prostate cancer: Recommendations of the RTOG-ASTRO Phoenix Consensus Conference. Int J Radiat Oncol Biol Phys 2006;65:965–974.
- 13. Cristofanilli M, Budd T, Ellis MJ, Stopeck A, Matera J, Miller MC et al. Circulating tumor cells, disease progresión, and survival in metastatic breast cancer. N Engl J Med 2004; 351:781-91.
- 14. Shaffer DR, Leversha MA, Danila DC, Lin O, Gonzalez-Espinoza R, Gu B et al. Circulating tumor cell analysis in patients with progresive castration-resistant prostate cancer. Clin Cancer Res 2007; 13(7):2023-29.
- 15. Almudena Zapatero, Mario A. López, Alicia Marín, Ricardo Mínguez, Feliciano García-Vicente. Dose-escalation with three-dimensional conformal radiotherapy for prostate cancer. Is more dose really better in high-risk patients treated with androgen deprivation? Clin Oncol 2006.18:600-607
- 16. Moreno JG, Miller MC, Gross S, Allard WJ, Gomella LG and Terstappen LW. Circulating tumor cells predict survival in patients with metastatic prostate cancer. Urology 2005; 65:713-18.
- 17. Fehm T, Sagalowsky A, Clifford E, Beitsch P, Saboorian H, Euhus D et al. Cytogenetic evidence that circulating epithelial cells in patients with carcinoma are malignant. Clin Cancer Res 2002; 8:2073-84.
- 18. Almudena Zapatero, Ricardo Mínguez, Santiago Nieto, Carmen Martín De Vidales, Feliciano García-Vicente. Post-Treatment Prostate Biopsies In The Era Of Three-Dimensional Conformal Radiotherapy. What Can They Teach Us? Eur Urol. 2009;55(902-910.
- 19. A. Zapatero, F. García-Vicente, C. Martín De Vidales, et al. Long-Term Results After High-Dose Radiotherapy And Adjuvant Hormones In Prostate Cancer: How Curable Is High-Risk Disease? IntJRadiatOncol BiolPhys2010 Oct 5. [Epub ahead of print] PMID:20932659[PubMed]

- 20. C. Olivier Gómeza y J. Carballido Rodríguez. Circulating tumor cells: Isolation, quantification, and relevante of their translation into clinical practice. actas urol esp. 2010;34(1):3-5.
- 21. Alix-Panabières C, Riethdorf S, Pantel K. Circulating tumor cells and bone marrow micrometastasis. Clin Cancer Res. 2008;14(16):5013-21.
- 22. Mocellin S, Keilholz U, Rossi CR, Nitti D. Circulating tumor cells: the 'leukemic phase' of solid cancers. Trends Mol Med. 2006;12(3):130-9.

## **RESPONSIBLE PARTY:**

Almudena Zapatero , MD PhD, PI - Promotor Hospital Universitario de la Princesa C/Diego de León, 62 Madrid 28006 E-mail: azapatero.hlpr@salud.madrid.org ID NUMBERS:

## **HEALTH AUTORITIES:**

Mª Rosario Ortiz de Urbina Barba Director Manager Fundación Investigación Biomédica IIS Hospital Universitario de la Princesa C/ Diego de León, 62 28006 Madrid

E-mail: mrosario.ortizurbina@salud.madrid.org